CLINICAL TRIAL: NCT00002210
Title: Phase II Study of the Safety, Tolerance, Pharmacokinetics, and Antiviral Effect of Delavirdine Mesylate (Rescriptor), in Combination With Nucleoside Reverse Transcriptase Inhibitors, in HIV-1-Infected Neonates, Infants, and Children
Brief Title: A Study of Delavirdine Mesylate in Combination With Other Anti-HIV Drugs in HIV-Infected Children and Babies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 228D; 0069
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-01

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Delavirdine; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Delavirdine

INTERVENTIONS:
Drug: Delavirdine mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give delavirdine mesylate (Rescriptor) plus two nucleoside reverse transcriptase inhibitors (NRTIs) to HIV-infected children and babies. This study also examines how the body processes Rescriptor when taken with 2 NRTIs.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Plasma HIV-1 levels greater than 10,000 copies/ml.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacia & Upjohn, Peapack, New Jersey, United States

REFERENCES:
- [Background] Willoughby R, Watson D, Welliver R. Early use of RESCRIPTOR (delavirdine) in children with HIV. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29 (abstract no 1995)